CLINICAL TRIAL: NCT06036810
Title: Engaging Patients in Decision Making: The Development and Pilot Testing of a Low Literacy Spanish Language Shared Medical Decision Tool for Ovarian Cancer Maintenance Therapy
Brief Title: Spanish Decision Tool for Ovarian Cancer Maintenance Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0539; NCI-2023-07034 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Phase 1 (Experimental): Pre-testing and cognitive interviews for the Decision Support Tool
  Interventions: Other: Shared Medical Decision Tool; Behavioral: Engaging Patients in Decision Making; Behavioral: Literacy Spanish Language
- Study Phase 2 (Experimental): Usual Care (Control Group) or Participants utilize the Decision Support Tool with Provider guidance (Intervention Group).
  Interventions: Other: Shared Medical Decision Tool; Behavioral: Engaging Patients in Decision Making; Behavioral: Literacy Spanish Language

INTERVENTIONS:
Other: Shared Medical Decision Tool — standard of care
Behavioral: Engaging Patients in Decision Making — standard of care
Behavioral: Literacy Spanish Language — standard of care

SUMMARY:
To develop a shared decision-making (SDM) tool to help Spanish-speaking patients make decisions about their maintenance therapy

DETAILED DESCRIPTION:
Objectives:

* Create a low literacy version of a shared decision-making (SDM) tool for ovarian cancer maintenance therapy for Spanish speaking individuals.
* To explore the feasibility and acceptability of incorporating the SDM tool into routine clinical care for Spanish speaking individuals.
* To estimate the effectiveness of the SDM tool on quality of the decision making in patients with ovarian cancer who are making decisions about maintenance therapy through a pilot study.

ELIGIBILITY:
Study population: This study will enroll patients and clinical providers.

Inclusion criteria: Patients

• Eligible patients must be: 1) individuals ≥ 18 years with advanced stage high grade epithelial ovarian, fallopian tube or primary peritoneal cancer who are receiving or have completed platinum-based chemotherapy for ovarian cancer and are potentially eligible to receive maintenance therapy; 2) able to understand, speak or read in Spanish.

Exclusion criteria: Patients

• Inability or unwillingness to sign informed consent

Inclusion criteria: Clinicians

• Eligible clinicians will include: 1) MD Anderson gynecologic oncologists and advanced practice providers who practice at the Houston Area Locations (HALs), MD Anderson Cancer Center, or our county safety net hospital, The Harris Health System (LBJ Hospital).

Exclusion criteria: Clinicians

• Inability or unwillingness to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Decision Regret Scale questionnaire | through study completion; an average of 2 year.
  This scale measures decisional regret related to health care decisions at a specific point in time. This tool consists of 5 questions answered on a Likert scale (1="Strongly agree" to 5="Strongly disagree").

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Meyer, Meyer, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org